CLINICAL TRIAL: NCT00865592
Title: An Open Label, Multi-Center, Long-Term Extension Study to Evaluate the Safety of PHX1149T/Dutogliptin in Subjects With Type 2 Diabetes Mellitus
Brief Title: Long-term Study to Evaluate the Safety of Dutogliptin/PHX1149T in Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Phenomix (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Hans-Peter Guler, MD, Phenomix
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHX1149-PROT300E
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes Mellitus; Type 2 Diabetes
Keywords: diabetes; DPP4 inhibitor; dutogliptin; PHX1149
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dutogliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dutogliptin — dutogliptin 400 mg, once daily tablet
  Other Names: PHX1149T; PHX1149; dutogliptin tartrate

SUMMARY:
The purpose of this study is to demonstrate that dutogliptin/PHX1149T is safe and tolerable.

DETAILED DESCRIPTION:
In this study, open-label dutogliptin/PHX1149T will be offered to subjects who complete a Phase 3 core protocol and wish to continue treatment with dutogliptin. This will allow for the collection of long-term safety data and will also demonstrate long-term effects on HbA1c and fasting blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Completion of all required visits of a qualifying Phase 3 core protocol (e.g., Visit 8/Day 196 of PHX1149-PROT301)
* Current treatment of Type 2 diabetes mellitus as in PHX1149-PROT301

Exclusion Criteria:

* Except for Type 2 diabetes, any other uncontrolled, serious pulmonary, cardiovascular, hematologic, renal, gastrointestinal, endocrine, neurological, proliferative, immunosuppressive, psychiatric, or urogenital disorder; or diseases of skin and its appendages, the eyes, ears, nose, or throat
* Any condition, disease, disorder or clinically relevant laboratory abnormality which, in the opinion of the investigator, would jeopardize the patient's appropriate participation in this study or obscure the effects of treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-01 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
To demonstrate safety and tolerability of dutogliptin | Two years

SECONDARY OUTCOMES:
To demonstrate maintenance or lowering of HbA1c | Two years
To demonstrate maintenance or lowering of fasting blood glucose | Two years

CONTACTS AND LOCATIONS:
Locations (68):
- United States (13):
  - Norwalk, California
  - Orange, California
  - Santa Ana, California
  - Daytona Beach, Florida
  - Kissimmee, Florida
  - Atlanta, Georgia
  - Phenomix Investigational Site 663, Honolulu, Hawaii
  - Brockton, Massachusetts
  - St Louis, Missouri
  - Cincinnati, Ohio
  - El Paso, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
- Argentina (6):
  - Phenomix Investigational Site 103, Buenos Aires
  - Phenomix Investigational Site 110, Buenos Aires
  - Phenomix Investigational Site 111, Buenos Aires
  - Phenomix Investigational Site 106, Caba
  - Phenomix Investigational Site 112, Corrientes
  - Phenomix Investigational Site 102, Paraná
- India (9):
  - Bangalore, Karnataka
  - Chennai, Tamil Nadu
  - Gulbarga, Karnataka
  - Hyderabad, Andhara Pradesh
  - Mumbai, Maharashtra
  - Nagpur, Maharashtra
  - Nashik, Maharashtra
  - Navi Mumbai, Maharashtra
  - Pune, Maharashtra
- Malaysia (6):
  - Phenomix Investigational Site 403, Kuching, Sarawak
  - Kelantan
  - Kuala Lumpur
  - Perak
  - Phenomix Investigational Site 404, Putrajaya
  - Sarawak
- Peru (6):
  - Phenomix Investigational Site 604, Arequipa
  - Phenomix Investigational Site 606, Lambayeque
  - Phenomix Investigational Site 600, Lima
  - Phenomix Investigational Site 601, Lima
  - Phenomix Investigational Site 602, Lima
  - Phenomix Investigational Site 609, Lima
- Philippines (4):
  - Phenomix Investigational Site 703, Cebu City
  - Manila, NCR
  - Quezon City, NCR
  - San Juan, NCR
- Romania (9):
  - Phenomix Investigational Site 802, Brasov
  - Phenomix Investigational Site 806, Brasov
  - Phenomix Investigational Site 800, Bucharest
  - Phenomix Investigational Site 803, Bucharest
  - Phenomix Investigational Site 805, Bucharest
  - Phenomix Investigational Site 807, Bucharest
  - Phenomix Investigational Site 804, Galati
  - Phenomix Investigational Site 801, Ploieşti
  - Phenomix Investigational Site 808, Sibiu
- Ukraine (15):
  - Phenomix Investigational Site 551, Ivano-Frankivsk
  - Phenomix Investigational Site 550, Kharkiv
  - Phenomix Investigational Site 557, Kharkiv
  - Phenomix Investigational Site 564, Kharkiv
  - Phenomix Investigational Site 555, Kiev
  - Phenomix Investigational Site 556, Kiev
  - Phenomix Investigational Site 562, Kiev
  - Phenomix Investigational Site 563, Kiev
  - Phenomix Investigational Site 554, Kylv
  - Phenomix Investigational Site 565, Lutsk
  - Phenomix Investigational Site 553, Lviv
  - Phenomix Investigational Site 561, Poltava
  - Phenomix Investigational Site 560, Simferopol
  - Phenomix Investigational Site 559, Vinnitsa
  - Phenomix Investigational Site 552, Zaporzhzhia